CLINICAL TRIAL: NCT01762540
Title: Glucocorticoid Induced Inhibition of IGF-I Activity: Exploring Underlying Mechanisms.
Brief Title: Glucocorticoid Induced Whole Body Catabolisme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: The Ministry of Science, Technology and Innovation, Denmark (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GK_nilani_2012
Record Dates: First submitted 2013-01-03; First posted 2013-01-07 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Whole Body Catabolisme Induced by Glucocorticoids
Keywords: Protein breakdown; Insulin resistance; Glucose intolerance; Lipolysis
MeSH Terms: conditions — Insulin Resistance; Glucose Intolerance | interventions — Glucocorticoids; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Calcium supplement (Placebo Comparator): Capsule with tablet of calclium supplement
  Interventions: Drug: Calcium Supplement
- Glucocorticoids (Active Comparator): Capsule with tablet of Prednisolone 37,5mg
  Interventions: Drug: Glucocorticoids

INTERVENTIONS:
Drug: Glucocorticoids — Prednisolone 37.5 mg x1 for 5 days
  Other Names: Prednisolone
  Arms: Glucocorticoids
Drug: Calcium Supplement — Placebo
  Other Names: Placebo
  Arms: Calcium supplement

SUMMARY:
The main purpose of the trial is to advance our knowledge on the possible mechanism underlying the catabolic effects of long-term treatment with glucocorticoid.

DETAILED DESCRIPTION:
Long-term treatment with glucocorticoid induces a general state of catabolism and increases insulin resistance. The underlying mechanisms are insufficiently characterized, however glucocorticoid induced changes of Growth Hormone (GH) and the Insulin-like growth factor I (IGF-I) appear to be of outmost importance.

We wish to investigate the mechanism behind glucocorticoid induced catabolism and insulin resistance.

More specific we wish to investigate:

* Whether glucocorticoid induces IGF-I inhibiting substances in serum or interstitial fluid that block the ability of IGF-I to phosphorylate its receptor in vitro
* Whether glucocorticoid inhibits intracellular IGF-I and insulin signaling in vitro and in vivo
* The mechanisms by which growth hormone counteracts the CG-mediated inhibition of IGF-I action

ELIGIBILITY:
Inclusion Criteria:

* signed and dated informed consent
* healthy subjects
* sex: male
* age 20-30 years
* BMI 19-26 kg/m2
* normal HbA1c

Exclusion Criteria:

* suspected og known allergy to the trial drug or similar medications.
* known current illness including diabetes mellitus, ischemic heart disease or cardiac arrhythmia.
* Daily drug intake (excluding Over-the-Counter medicines).
* Known or previous mental illness
* Current participation or previous participation in experiments using ionizing radiation for a year prior to inclusion in this study.
* Participation in a larger X-ray examinations in trial period.

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Insulin-like Growth Factor (IGF)-I profiles of subjects before and after prednisolone-treatment. | day 1, 3 and 5
  Blood-test before (day 1) during (day 3) and at the end (day 5) of placebo/prednisolone treatment.

SECONDARY OUTCOMES:
Intracellular signaling of IGF-I under the influence/abscence of prednisolone. | day 5
  Tissue biopsy on day 5.
Insulin sensitivity under the influence/abscence of prednisolone. | Day 5
  Hyperinsulinemic euglycemic clamp on day 5.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Frystyk, Professor, Principal Investigator — Medical Research Laboratory, Clinical institute of Medicine, Aarhus University Hospital
Locations (1):
- Medical Research Laboratory, Clinical Institute of Medicine, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Ramshanker N, Jessen N, Voss TS, Pedersen SB, Jorgensen JOL, Nielsen TS, Frystyk J, Moller N. Effects of short-term prednisolone treatment on indices of lipolysis and lipase signaling in abdominal adipose tissue in healthy humans. Metabolism. 2019 Oct;99:1-10. doi: 10.1016/j.metabol.2019.06.013. Epub 2019 Jun 29. PMID 31260678
- [Derived] Ramshanker N, Aagaard M, Hjortebjerg R, Voss TS, Moller N, Jorgensen JOL, Jessen N, Bjerring P, Magnusson NE, Bjerre M, Oxvig C, Frystyk J. Effects of Prednisolone on Serum and Tissue Fluid IGF-I Receptor Activation and Post-Receptor Signaling in Humans. J Clin Endocrinol Metab. 2017 Nov 1;102(11):4031-4040. doi: 10.1210/jc.2017-00696. PMID 28945869